CLINICAL TRIAL: NCT00616720
Title: Randomized Phase II Trial of Dendritic Cell-Based Idiotype Vaccination With Adjuvant Cytokines for Plateau Phase and Post-Transplant Multiple Myeloma
Brief Title: Interferon-gamma or Aldesleukin and Vaccine Therapy in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Martha Q. Lacy, M.D., Mayo Clinic Cancer Center
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000582566; P30CA015083 (NIH); 998003 (Other: Mayo Clinic Cancer Center); 789-99 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-02-14; First posted 2008-02-15 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — aldesleukin; Interferon-gamma; Polymerase Chain Reaction; Reverse Transcriptase Polymerase Chain Reaction; Flow Cytometry

INTERVENTIONS:
Biological: aldesleukin
Biological: idiotype-pulsed autologous dendritic cell vaccine APC8020
Biological: recombinant interferon gamma
Genetic: polymerase chain reaction
Genetic: reverse transcriptase-polymerase chain reaction
Other: flow cytometry
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Biological therapies, such as interferon-gamma and aldesleukin, may stimulate the immune system in different ways and stop cancer cells from growing. Vaccines made from a person's white blood cells may help the body build an effective immune response to kill cancer cells. Giving biological therapy together with vaccine therapy may kill more cancer cells.

PURPOSE: This randomized phase II trial is studying how well giving aldesleukin or interferon gamma together with vaccine therapy works in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the clinical benefit in patients with plateau phase multiple myeloma treated with interferon-gamma vs aldesleukin in combination with idiotype-pulsed autologous dendritic cell vaccine APC8020.
* To describe response rates in patients who are in plateau phase status post-chemotherapy or status post-peripheral blood cell transplantation treated with this regimen.

Secondary

* To obtain data regarding the ability of this approach to produce an anti-idiotypic immunologic response.
* To obtain information about the effects of interferon-gamma and aldesleukin on the number, function, and activation state of immune effector-cells including T-cells and B-cells.
* To perform detailed analyses of lymphocyte phenotypes and T-cell repertoires before and after idiotype-pulsed autologous dendritic cell vaccine APC8020.

OUTLINE: Patients are stratified according to gender (male vs female) and prior treatment (post-chemotherapy vs post-peripheral blood stem cell transplantation). Patients are randomized to 1 of 2 arms.

In both arms, patients undergo apheresis for collection of peripheral blood mononuclear cells for generation of dendritic cells (DC) on days 0, 14, and 28. APC8020 is generated by loading DC with immunoglobulin idiotype prepared from the patient's serum.

* Arm I: Patients receive interferon-gamma subcutaneously (SC) once daily on days 1-5, 15-20, and 29-34 and idiotype-pulsed autologous dendritic cell vaccine APC8020 IV over 30-minutes on days 2, 16, and 30.
* Arm II: Patients receive aldesleukin SC once daily days 1-5, 15-20, and 29-34 and idiotype-pulsed autologous dendritic cell vaccine APC8020 as in arm I.

In both arms, treatment continues in the absence of disease progression.

Peripheral blood samples are collected at baseline and on day 5 of courses 1 and 4 for cytokine immunomodulatory studies, including immunophenotyping for lymphocyte phenotypic markers (CD69, CD40L, CD25, CD30, CD71, CDW137, CD134, and HLADR) by flow cytometry and immunofluorescence; T-cell spectratyping by PCR and RT-PCR; T-cell proliferation to idiotype protein; and CTL and T-helper response by flow cytometry.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma
* Plateau phase multiple myeloma (status post chemotherapy or status post-peripheral blood cell transplantation), meeting the following criteria:

  * Serum and urine monoclonal (M) protein values must be stable (< 20% variation) or must have disappeared
  * Serum M protein < 1 g/dL, and 1 of the following:

    * Quantifiable serum M protein
    * Adequate serum sample stored in Transfusion Medicine under IRB protocol #698-98
  * Urine M protein < 200 mg/24 hours by electrophoresis on 2 separate occasions for a period of ≥ 4 weeks
* Serum M protein spike ≤ 2.0 g/dL
* No progressive disease after prior autologous stem cell transplantation or chemotherapy
* No non-secretory or light chain myeloma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 6 months
* WBC ≥ 1,500/μL
* Platelet count ≥ 50,000/μL
* Total bilirubin ≤ 5 times upper limit of normal
* Creatinine ≤ 5.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must have adequate venous access for apheresis
* No uncontrolled cardiac disease
* No uncontrolled infection
* No illness or condition which, in the opinion of the investigator, may affect safety of treatment or evaluation of any of the study's endpoints

PRIOR CONCURRENT THERAPY:

* Recovered from all prior therapy
* More than 4 weeks since prior standard-dose chemotherapy, radiotherapy, or immunotherapy
* More than 3 months since prior high-dose chemotherapy with stem cell transplantation
* No concurrent corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2001-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Confirmed response (i.e., clinical or immunological)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Q. Lacy, MD, Study Chair — Mayo Clinic